CLINICAL TRIAL: NCT04828616
Title: An Open-label, Multicentre, Phase II Study of DP303c Injection in Patients With HER2-expressing Advanced Ovarian Cancer
Brief Title: Study of DP303c Injection in Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1501-CSP-002
Record Dates: First submitted 2021-03-28; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DP303c injection (Experimental): Part1:Patients with HER2-expressing advanced ovarian cancer will be treated with DP303c injection at 2.0 mg/kg or 3.0 mg/kg every 3 weeks (Q3W) to determine the recommended phase 2 dose (RP2D).
  Part2a:Patients with HER2-overexpressing advanced ovarian cancer will be treated with DP303c injection at RP2D.
  Part2b:Patients with HER2-lowexpressing advanced ovarian cancer will be treated with DP303c injection at RP2D.
  Interventions: Drug: DP303c injection

INTERVENTIONS:
Drug: DP303c injection — DP303c injection, every 3 weeks (Q3W)
  Other Names: DP303c

SUMMARY:
This study is an open-label, multicentre, phase II study to evaluate the efficacy and safety of of DP303c injection in patients with HER2-expressing advanced ovarian cancer.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II study of DP303c injection in patients with HER2-expressing advanced ovarian cancer with two parts. In part 1, patients will be treated with DP303c injection at two dose levels (2.0 mg/kg or 3.0 mg/kg) every 3 weeks to determine the recommended phase 2 dose (RP2D). Once the RP2D has been established in part 1, patients will be enrolled into 2 cohorts in part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent.
2. Aged 18 to 75 years, female.
3. Histologically or cytologically confirmed epithelial ovarian cancer, carcinoma tubae, or primary peritoneal carcinoma.
4. Patients have previously received platinum-containing chemotherapy.
5. Patients must provide tissue samples that are certified as qualified by the central laboratory, and the HER2 status of the tissue samples is determined by the central laboratory:Part1: HER2 overexpressing: IHC 2+ or IHC 3+; Part2a: HER2 overexpressing: IHC 2+ or IHC 3+; Part2b: HER2 low expressing: IHC1+;
6. The Eastern Cooperative Oncology Group (ECOG) score is 0 to 2, and life expectancy ≥ 3 months.
7. At least one measurable lesion at baseline per RECIST v1.1.
8. The function of major organs must meet the following criteria within 7 days before enrollment (Have not received blood transfusion, EPO, G-CSF or other medical supportive treatment within 14 days before the first dose of study drug):

   Absolute neutrophil count (ANC) ≥1.5×109/L, Platelet ≥100×109 /L; Hemoglobin ≥90 g/L or ≥5.6 mmol/L; International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN; Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN; Creatinine clearance rate ≥30 mL/min (Calculated by Cockcroft-Gualt formula); Total bilirubin ≤1.5×ULN or ≤3×ULN for patients with Gilbert's syndrome or liver metastasis: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5×ULN or ≤5×ULN for patients with liver metastasis:
9. Female patient of childbearing age must agree to take adequate contraceptive measures during the entire study period and through at least 6 months after the last dose of study drug. Women of childbearing age must have a negative pregnancy test within 7 days before study entry.
10. Patients will be able to communicate well with the investigator, understand and comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Has not recovered from adverse reactions caused by previous anti-tumor treatments to ≤ grade 1 or baseline (refer to NCI CTCAE 5.0), except for alopecia, pigmentation and other toxicity judged no safety risk by the investigator .
3. Patients who have previously received trastuzumab or trastuzumab analogues that have related toxicity, resulting in permanent discontinuation.
4. Patients with allergic history or delayed allergic reaction to any components (trastuzumab analogues, MMAE, sodium citrate dihydrate, citrate monohydrate, polysorbate 20 and sucrose, etc.) of DP303c.
5. Patients with brain or pia mater metastasis, except for patients with central nervous system (CNS) metastases in the following conditions: untreated but asymptomatic, or progression-free status in imaging evidence for at least 4 weeks after treatment and not requiring hormone therapy for at least 4 weeks.
6. Chemotherapy, radiotherapy, biotherapy, targeted therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first dose of study drug, 6 weeks for nitrosourea (such as carmustine, lomustine, etc.) or mitomycin C, 5 half-lives for oral fluorouracil and small molecule targeted drugs, 2 weeks for endocrine therapy and Chinese medicine treatment with anti-tumor indications; or local palliative radiotherapy for bone metastasis and pain relief within 2 weeks.
7. People who currently have corneal diseases that require medication or surgical intervention, or have a history of serious corneal diseases, or are unwilling to stop wearing contact lenses during the study.
8. History of any other malignant tumors within five years (except for skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, local prostate cancer, cervical cancer in situ, stage I ductal carcinoma in situ and stage I grade 1 endometrial carcinoma that have been radically removed and have not recurred; breast cancer with no recurrence for more than 3 years after radical operation).
9. History of (non-infectious) interstitial lung disease (ILD)/pulmonary disease that required steroids, or current ILD/pulmonary disease, or suspected ILD/ pulmonary disease that cannot be excluded by imaging examination; except for patients with radiation pneumonitis without clinical symptoms after 3 months of radiotherapy.
10. Patients with dyspnea at rest induced by complications of advanced malignant tumors or need for continuous oxygen therapy.
11. Patients with complete intestinal obstruction, or pleural effusions or ascites that are difficult to control within 4 weeks before entry (the frequency of percutaneous drainage is more than twice a week, or continuous drainage daily volume is ≥ 1000 mL).
12. Patients with serious cardiovascular and cerebrovascular diseases, including but not limited to:

    * Uncontrolled angina, congestive heart failure (NYHA III-IV), myocardial infarction or severe arrhythmia within 6 months before enrollment;
    * Left ventricular ejection fraction (LVEF) <50% or lower limit of normal in echocardiogram (ECHO) or multi-gate detection scan (MUGA);
    * Average adjusted QT interval prolongation >470 ms, QT interval corrected by Fridericia's formula (QTcF).
13. The cumulative amount of previous exposure to anthracyclines has reached the following doses: doxorubicin or liposomal doxorubicin>500 mg/m2; epirubicin>900 mg/m2; mitoxantrone>120 mg/m2; Others (liposomal doxorubicin or other anthracyclines is equivalent to a dose of > 500 mg/m2 adriamycin); if more than one anthracycline is used, the cumulative dose is equivalent to a total dose of >500 mg/m2 adriamycin.
14. Peripheral neuropathy ≥grade 2 before entry (NCI CTCAE 5.0).
15. Uncontrollable electrolyte imbalances include hypokalemia, hypocalcemia or hypomagnesemia (refer to NCI CTCAE 5.0, ≥2 grade).
16. HIV positive, or syphilis infection requiring systematic treatment.
17. Patients with active hepatitis B or C (HBsAg positive, with HBV DNA positive, and the ALT continues to be higher than the upper limit of normal, without other causes of ALT elevation; HCVAb positive with HCV RNA higher than the upper limit of normal).
18. Patients have used strong CYP3A4 inhibitors or CYP3A4 strong inducers with a washout period less than 28 days or 5 half-lives (whichever is shorter) before the first dose of the study drug.
19. Patients underwent major surgery within 4 weeks and did not fully recover before the first dose of study drug.
20. Patients have received other clinical trial drugs within 4 weeks before the first dose of study drug.
21. Have previously received antibody drug conjugate targeting HER2.
22. Patients with any mental or cognitive impairment that may restrict their understanding and implementation of the informed consent form.
23. Other serious or uncontrollable diseases or conditions that may affect the evaluation of the primary endpoint or the investigator believes that participation in this study may bring risks to the patient.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Through study completion, an average of 3 year
  Objective Response Rate is defined as the percentage of patients with a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
PFS | Through study completion, an average of 3 year
  Progression Free Survival
OS | From the enrollment to the death of last subject or the end of the clinical trial (assessed up to 36 months)
  Overall Survival
Duration of Response (DoR) | Through study completion, an average of 3 year
  To preliminarily evaluate DoR in patients with advanced solid tumors
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Through study completion, an average of 3 year
  The drug safety will be assessed by investigator(s) according to NCI-CTCAE v5.0.
Maximum concentration (Cmax) of DP303c | Part1:Cycle 1 Day 1, Cycle 1 Day 8,Cycle 1 Day 15, Cycle 2 Day 1 ,Cycle 2 Day 15,Cycle 3 Day 1and Cycle 5 Day 1;Part2:Cycle 1 Day 1, Cycle 1 Day 8,Cycle 1 Day 15, Cycle 2 Day 1 ,Cycle 2 Day 15; predose. A cycle is 21 days
  The pharmacokinetics(PK) profile of DP303c
Time of peak plasma concentration (Tmax) | Part1:Cycle 1 Day 1, Cycle 1 Day 8,Cycle 1 Day 15, Cycle 2 Day 1 ,Cycle 2 Day 15,Cycle 3 Day 1and Cycle 5 Day 1;Part2:Cycle 1 Day 1, Cycle 1 Day 8,Cycle 1 Day 15, Cycle 2 Day 1 ,Cycle 2 Day 15; predose. A cycle is 21 days
  The pharmacokinetics(PK) profile of DP303c
Area under the plasma concentration time curve (AUC) of DP303c | Part1:Cycle 1 Day 1, Cycle 1 Day 8,Cycle 1 Day 15, Cycle 2 Day 1 ,Cycle 2 Day 15,Cycle 3 Day 1and Cycle 5 Day 1;Part2:Cycle 1 Day 1, Cycle 1 Day 8,Cycle 1 Day 15, Cycle 2 Day 1 ,Cycle 2 Day 15; predose. A cycle is 21 days
  The pharmacokinetics(PK) profile of DP303c
Immunogenicity (anti-drug antibody ADA) | Through study completion, an average of 3 year
  Percentage of patients producing detectable ADA.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China